CLINICAL TRIAL: NCT05199298
Title: The Effect of Mandala Activity-Based Breastfeeding Program on Breastfeeding Self-Efficacy and Maternal-Infant Attachment of Primiparous Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Çiğdem Sarı Öztürk, Dr. Cigdem Sarı Ozturk-Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CSOzturk
Record Dates: First submitted 2022-01-01; First posted 2022-01-20 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Breastfeeding; ART; Self Efficacy; Maternal-Fetal Relations
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Mandala Activity-Based Breastfeeding Program" (Experimental): The group receiving Mandala Activity-Based Breastfeeding Program
  Interventions: Other: "Mandala Activity-Based Breastfeeding Program"
- Control group (No Intervention): the group that did not receive any training/initiative

INTERVENTIONS:
Other: "Mandala Activity-Based Breastfeeding Program" — Training modules for breastfeeding and Maternal -infant attachment will be implemented with pregnant women in the study group at 32-36 weeks of gestation. The training will be explained by the researchers by shooting a video. In addition, for each week, mandala drawings will be videotaped by the researcher who received mindfulness-based art therapy training and will be sent to the Whatsapp accounts of the pregnant women. t 36 weeks of gestation, the Prenatal Attachment Scale and Spielberger State Anxiety Inventories will be sent to mothers as Google forms. The mother will be called 24 hours after the birth and the situation of having a problem with breastfeeding will be determined. In the first week, in the first and second months after the birth, questionnaire forms and online questionnaires will be applied to the mothers, apart from the follow-up and counseling in the postpartum 2nd month, the posttests of the scales
  Arms: "Mandala Activity-Based Breastfeeding Program"

SUMMARY:
This study will be conducted to determine the effect of breastfeeding program integrated with art therapy such as mandala painting on postpartum breastfeeding self-efficacy, breastfeeding rates, and mother-infant attachment of primiparous mothers.

Training on breastfeeding and mother-baby bonding and mandala drawings supporting the training will be sent online to primiparous pregnant women who are at 32-36 weeks of gestation and agree to participate in the study. Telephone follow-up and counseling will continue in the postpartum period. In the postpartum period, follow-up and counseling will continue until the second month.

DETAILED DESCRIPTION:
In this study, a mandala-based breastfeeding program will be applied to primiparous mothers at 32-36 weeks of gestation. The study will be conducted to determine the effect of mandala-based breastfeeding programs on postpartum breastfeeding self-efficacy, breastfeeding rates, and maternal-infant attachment of primiparous mothers. Training on breastfeeding and mother-baby bonding and mandala drawings supporting training will be sent online to primiparous pregnant women who are at 32-36 weeks of gestation and agree to participate in the study. The study is planned to be conducted with 72 pregnant women (intervention group=36, control group=36). Telephone follow-up and counseling will continue in the postpartum period. In the postpartum period, follow-up and counseling will continue until the second month.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous pregnancy,
* Being at 32-33 weeks of gestation,
* Being over 18 years old,
* To be at least a primary school graduate,
* Owning a phone,
* Having internet access at home or at work,
* Using the internet,
* Being able to speak Turkish,
* Mothers who agreed to participate in the study

For infants;

* Born at 37-42 weeks of gestation,
* Birth weight between 2500-4000 g,
* Infants without any health problems or congenital anomalies were included in the study.

Exclusion Criteria:

* pregnant women and infants with health problems

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
The Spielberger State-Trait Anxiety Inventory (STAI) | Change from Baseline level of Spielberger State-Trait Anxiety to 2 months (change is being assessed)]
  The scale is a 20-item self-report measure of anxiety using a 4-point Likert-type scale (from 0 to 3 points) for each item. The total score obtained from the scale varies between 20 and 80. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety.
Maternal Attachment Scale | Change from Baseline level of Maternal Attachment Scale at 2 months (change is being assessed)].
  The scale consists of 26 statements and is a four-point Likert type. High score indicates that maternal attachment is high. The scores obtained from the scale range from a minimum of 26 to a maximum of 104 points
Postnatal Breastfeeding Self-Efficacy Scale | Change from Baseline level of Postnatal Breastfeeding Self-Efficacy Scale at 2 months (change is being assessed)].
  The scale is 5-point Likert type and consists of 14 items. The lowest score that can be obtained from the scale is 14, and the highest score is 70. A higher score means higher breastfeeding self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Sari Ozturk C, Demir K. The Effect of Mandala Activity and Technology-Based Breastfeeding Program on Breastfeeding Self-Efficacy and Mother-Infant Attachment of Primiparous Women: A Randomized Controlled Study. J Med Syst. 2023 Apr 1;47(1):44. doi: 10.1007/s10916-023-01942-3. PMID 37004692